CLINICAL TRIAL: NCT07357324
Title: A Clinical Observation Study of a Chinese Patent Medicine Combined With Tamsulosin in Improving Sleep and Nocturia Symptoms After Enucleation of the Prostate
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-2025-144
Record Dates: First submitted 2025-12-11; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Benign Prostatic Hyperplasia; Nocturia Associated With Nocturnal Polyuria
Keywords: Benign Prostatic Hyperplasia; Transurethral Holmium Laser Enucleation of Prostate; Tamsulosin; Lingze Tablets
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

STUDY DESIGN:
Intervention Model Description: Two-arm parallel randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: This is a single-blind study. Due to the different dosing regimens between the two groups (tamsulosin once daily vs. tamsulosin once daily plus Lingze tablets three times daily), it is not possible to blind participants or care providers. However, the outcomes assessors responsible for collecting questionnaire data (IPSS, PSQI, HAMA) and urodynamic measurements will be blinded to group allocation. Additionally, the statistician/data analyst will remain blinded to treatment assignments during data processing and analysis to minimize bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tamsulosin Monotherapy Group (Active Comparator): Participants in this arm will receive tamsulosin hydrochloride sustained-release capsules (0.2 mg) orally once daily at bedtime for 8 weeks. This represents the standard postoperative pharmacological treatment following transurethral holmium laser enucleation of the prostate. The medication (National Drug Approval Number: H20000681) is manufactured by Jiangsu Hengrui Medicine Co., Ltd. Participants will be instructed to take the capsule with water and avoid crushing or chewing it. Regular monitoring for adverse events, medication adherence, and urinary/sleep symptom progression will be conducted at baseline, Week 4, and Week 8 visits.
  Interventions: Drug: Tamsulosin Hydrochloride Sustained-Release Capsules
- Lingze Tablets Combined with Tamsulosin Group (Experimental): Participants in this arm will receive combination therapy consisting of Lingze tablets plus tamsulosin hydrochloride sustained-release capsules for 8 weeks. Lingze tablets (National Drug Approval Number: Z20110050), manufactured by Zhejiang Conba Pharmaceutical Co., Ltd., will be administered orally at a dose of 4 tablets three times daily. Tamsulosin hydrochloride sustained-release capsules (0.2 mg) will be administered orally once daily at bedtime. This experimental intervention aims to evaluate whether the addition of Lingze tablets, a traditional Chinese patent medicine with kidney-tonifying and dampness-clearing properties, to standard tamsulosin therapy provides superior improvement in postoperative nocturia and sleep quality compared to tamsulosin monotherapy. Participants will be monitored for medication adherence, adverse events, and clinical outcomes at baseline, Week 4, and Week 8 visits.
  Interventions: Drug: Tamsulosin Hydrochloride Sustained-Release Capsules; Drug: Lingze Tablets

INTERVENTIONS:
Drug: Tamsulosin Hydrochloride Sustained-Release Capsules — Tamsulosin is an alpha-1 adrenergic receptor antagonist used as standard therapy to relieve lower urinary tract symptoms by relaxing the smooth muscle of the bladder neck and prostate. This study uses 0.2 mg sustained-release capsules administered orally once daily at bedtime for 8 weeks. The medication (National Drug Approval Number: H20000681) is manufactured by Jiangsu Hengrui Medicine Co., Ltd. It is administered to participants in both the control arm (monotherapy) and the experimental arm (combination therapy).
  Other Names: Tamsulosin; α1-adrenergic receptor antagonist
Drug: Lingze Tablets — Lingze tablets are a traditional Chinese patent medicine composed of herbal extracts including Rhizoma Alismatis, Poria, Radix Rehmanniae Preparata, Rhizoma Curculiginis, and Herba Epimedii. According to traditional Chinese medicine theory, it tonifies kidney qi, clears dampness and heat, and promotes blood circulation to alleviate urinary symptoms. In this study, it is administered orally at 4 tablets three times daily for 8 weeks, in combination with tamsulosin, to participants in the experimental arm only. The product (National Drug Approval Number: Z20110050) is manufactured by Zhejiang Conba Pharmaceutical Co., Ltd.
  Arms: Lingze Tablets Combined with Tamsulosin Group

SUMMARY:
This study will test whether a traditional Chinese medicine called Lingze tablets, when added to the standard drug tamsulosin, can better improve sleep and nighttime urination problems in men after prostate surgery.

Who can participate? Men aged 50 years or older who have had transurethral holmium laser enucleation of the prostate (a minimally invasive surgery for enlarged prostate) and continue to have bothersome nighttime urination (at least 2 times per night) and other urinary symptoms may be eligible.

Who cannot participate? Men who cannot tolerate the study medications, have severe cancer, serious organ failure, or have conditions that prevent them from understanding or following the study requirements.

What will participants do?

About 136 participants will be randomly assigned (by chance, like a coin flip) to one of two groups:

Group 1: Take tamsulosin sustained-release capsule once daily for 8 weeks Group 2: Take tamsulosin sustained-release capsule once daily PLUS Lingze tablets (4 tablets, three times daily) for 8 weeks Participants will visit the hospital clinic at the start of the study, at 4 weeks, and at 8 weeks for assessments.

What will be measured?

Researchers will measure:

How many times you wake up at night to urinate Overall sleep quality using standard questionnaires Prostate symptom scores and quality of life Urine flow tests (non-invasive) Anxiety levels Any side effects or adverse events from the medications Why is this study important? Many men continue to have nighttime urination and poor sleep even after prostate surgery, which can greatly reduce quality of life. This study will help determine if combining Lingze tablets with standard treatment provides better relief than standard treatment alone.

Risks and Benefits:

Potential benefits: Improved sleep, fewer nighttime bathroom trips, better urinary symptoms, and enhanced quality of life.

Potential risks: Possible side effects include dizziness, headache, nausea, or stomach upset from the medications. All participants will be closely monitored for any problems and can contact the study team 24/7 with concerns.

Privacy:

All personal and medical information will be kept confidential and used only for research purposes in accordance with hospital and national regulations.

DETAILED DESCRIPTION:
This study is designed to test whether adding a traditional Chinese medicine called Lingze tablets to the standard treatment (tamsulosin) can better relieve nighttime urination and sleep problems in men who have recently undergone a minimally invasive prostate surgery.

Why This Study Is Needed Many men develop an enlarged prostate (benign prostatic hyperplasia, or BPH) as they age, which can cause bothersome urinary symptoms. The standard surgical treatment is transurethral holmium laser enucleation of the prostate, a procedure that removes part of the prostate to improve urine flow. While this surgery is effective, up to half of men continue to experience significant urinary symptoms afterward, particularly needing to wake up frequently at night to urinate (nocturia). Poor sleep due to nocturia leads to daytime fatigue, reduced quality of life, and emotional distress. Current medications like tamsulosin (which relaxes the bladder and prostate muscles) help some men but don't fully resolve symptoms for everyone. Lingze tablets are a Chinese patent medicine made from herbal ingredients that, according to traditional Chinese medicine theory, work by strengthening kidney function and clearing dampness and heat from the body. Previous small studies suggest Lingze tablets may help with urinary symptoms, but this has not been tested in men after prostate surgery or combined with standard treatment.

Study Design

This is a randomized, parallel-group, controlled clinical trial meaning:

Randomized: Participants are assigned by chance (like flipping a coin) to one of two treatment groups. This helps ensure the groups are similar and the results are fair.

Parallel-group: Both groups are treated at the same time and followed for the same duration.

Controlled: One group receives the standard treatment alone, while the other receives standard treatment plus the study medication. This allows researchers to see if the combination is truly better.

Treatment Groups and Medications Group 1 (Control, about 68 participants): Takes one capsule (0.2 mg) of tamsulosin sustained-release orally once daily at bedtime for 8 weeks. This is the standard medication commonly prescribed after prostate surgery to help with urinary symptoms. The specific product is manufactured by Jiangsu Hengrui Medicine Co., Ltd. (National Drug Approval Number: H20000681).

Group 2 (Experimental, about 68 participants): Takes the same dose of tamsulosin once daily at bedtime PLUS Lingze tablets (4 tablets, three times daily) for 8 weeks. Lingze tablets are manufactured by Zhejiang Conba Pharmaceutical Co., Ltd. (National Drug Approval Number: Z20110050). Each Lingze tablet contains herbal extracts including Rhizoma Alismatis, Poria, Radix Rehmanniae Preparata, Rhizoma Curculiginis, and Herba Epimedii. The combination aims to both relax the urinary tract (tamsulosin) and address underlying imbalances that traditional Chinese medicine associates with urinary problems (Lingze).

All participants will receive standard postoperative care instructions, including guidance on diet, fluid intake, and activity levels.

Participant Journey: What to Expect

If you decide to participate, here is what will happen:

Visit 0 (Baseline, Week 0):

You will meet with the study doctor and nurse to review the study details and ask questions.

If you agree to participate, you will sign the informed consent form. The team will collect basic information about you (age, medical history, how long you've had symptoms, other health conditions).

You will complete several questionnaires that ask about your urinary symptoms, sleep quality, and anxiety levels (these take about 20-30 minutes total).

You will undergo a non-invasive urine flow test where you urinate into a special device that measures how fast and how much you urinate. This helps measure bladder function.

You will be randomly assigned to one of the two treatment groups and receive your first 4-week supply of medications with detailed instructions.

The research team will explain how to take the medications, what side effects to watch for, and how to contact them with any concerns (a 24-hour hotline will be provided).

Visit 1 (Week 4):

You will return to the clinic with your medication bottles so the team can check how well you have been taking the medications (adherence check).

You will complete the same questionnaires as at baseline to track any changes in your symptoms, sleep, and quality of life.

You will report any side effects or problems you have experienced. The doctor will answer your questions and provide health education about managing urinary symptoms.

You will receive your second 4-week supply of medications.

Visit 2 (Final Visit, Week 8):

You will return to the clinic for your final assessment. You will repeat all the questionnaires and the urine flow test. You will return all medication bottles for a final adherence check. The team will review your overall experience, any side effects, and your symptom improvement.

You will receive advice on continuing your treatment plan with your regular doctor after the study ends.

Throughout the 8-week period, you are encouraged to contact the study team at any time if you have questions, concerns about side effects, or any health issues. The team will also contact you by phone, text message, or email between visits as needed to check on your progress.

How We Will Measure Success: Outcome Measures

The study will evaluate several key areas:

Urinary Symptom Severity (IPSS): The International Prostate Symptom Score is a 7-question survey that asks how often you experience symptoms like incomplete emptying, frequent urination, weak stream, and nighttime urination. Each question is scored from 0 (not at all) to 5 (almost always), for a total score of 0-35. Lower scores mean fewer symptoms. This is the most common tool used worldwide to assess prostate-related urinary problems.

Quality of Life Impact (QOL): A single question asks: "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that?" You rate your answer from 0 (delighted) to 6 (terrible). This helps us understand how much your symptoms truly bother you.

Nighttime Urination (Nocturia): Specifically, we will count how many times you wake up each night to urinate. The IPSS questionnaire includes this as one item, but we will also track it separately as a primary focus of this study.

Sleep Quality (PSQI): The Pittsburgh Sleep Quality Index asks 19 questions about your sleep over the past month, covering 7 areas: sleep quality, how long it takes you to fall asleep, total sleep time, sleep efficiency (time in bed vs. time asleep), sleep disturbances (like waking up at night), use of sleep medications, and daytime sleepiness. Each area is scored 0-3, for a total score of 0-21. A lower score means better sleep quality. This is a well-validated tool used internationally.

Bladder Function (Urodynamic Parameters): We will perform simple, non-invasive tests:

Maximum Urine Flow Rate (Qmax): Measures the fastest speed of your urine stream (in milliliters per second). A higher number means better flow.

Average Urine Flow Rate (Qave): Measures the average speed throughout your urination.

Residual Urine Volume (RUV): Uses ultrasound to measure how much urine remains in your bladder after you urinate. Less residual urine means your bladder is emptying more completely.

Anxiety Level (HAMA): The Hamilton Anxiety Rating Scale includes 14 items about anxiety symptoms (like tension, fear, insomnia, muscle aches). Each item is rated from 0 (not present) to 4 (severe). The total score helps us understand if urinary and sleep problems are affecting your emotional health.

Safety and Side Effects: At every contact, we will ask about any health problems, symptoms, or concerns you have experienced. We will record details about any adverse events: what happened, when it started, how severe it was, how long it lasted, what was done about it, and what the outcome was. Common potential side effects from these medications include dizziness (especially when standing up), headache, nasal congestion, fatigue, nausea, or stomach discomfort. Most side effects are mild and temporary.

Sample Size and Statistics We calculated that we need 136 participants (68 in each group) to have enough statistical power to detect a meaningful difference between the two treatments. This calculation assumes that the combination therapy will reduce nighttime urination by at least 1 fewer episode per night compared to tamsulosin alone, with a 90% chance of detecting this difference if it truly exists. We added extra participants to account for an estimated 20% who might drop out or be lost to follow-up.

Data will be analyzed using SPSS 20.0 software. For continuous measures (like scores and urine flow rates), we will compare the average changes between groups using t-tests. For categorical data (like percentages of people with side effects), we will use chi-square tests. A p-value less than 0.05 will be considered statistically significant, meaning the difference is unlikely to be due to chance.

Quality Control and Data Integrity

To ensure reliable results, we will:

Verify that all participants meet strict inclusion and exclusion criteria before enrollment.

Use a random number table generated by computer to assign participants to groups, preventing any bias.

Check medication adherence at each visit by counting remaining pills and asking participants about missed doses.

Monitor for adverse events continuously and have a physician available 24/7 for urgent concerns.

Keep the data analysts "blinded" to which participant is in which group until the final analysis is complete, to prevent unconscious bias in interpreting results.

Use standardized, validated questionnaires and measurement techniques at all time points.

Privacy and Confidentiality All information collected about you will be kept strictly confidential. Your data will be assigned a unique study ID number, and your name and other direct identifiers will be stored separately in a password-protected database accessible only to essential study staff. Any information published or presented will not identify you personally. All data collection, storage, and analysis comply with hospital policies and national regulations protecting research participants.

Participation Rights

Your participation is completely voluntary. You have the right to:

Ask questions about the study at any time Refuse to participate without any penalty or loss of medical care Withdraw from the study at any time for any reason Receive a copy of your signed consent form Be informed of any new information that might affect your willingness to continue Contact Information

For questions about the study, your rights as a participant, or to report problems, you can contact:

Principal Investigator: Dr. Guangyi Huang 24-Hour Study Hotline: [To be provided at enrollment] Institutional Review Board: [Hospital Ethics Committee contact information will be provided] Results Sharing After the study is completed, we plan to publish the findings in a medical journal and present them at scientific conferences. A summary of results will be made available to all participants who request it.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 50 years or older
* History of transurethral holmium laser enucleation of the prostate (HoLEP)
* Nocturia frequency ≥2 times per night
* Documented bladder outlet obstruction
* Presence of postoperative urinary incontinence and urgency symptoms
* Ability to understand study procedures and provide written informed consent
* Willingness to complete all scheduled follow-up visits and assessments

Exclusion Criteria:

* Known hypersensitivity or intolerance to tamsulosin hydrochloride, Lingze tablets, or any component of these medications
* Active malignancy or severe cancer requiring treatment
* Cognitive impairment, psychiatric disorder, or language barrier that prevents understanding of study requirements or completion of questionnaires
* Severe multi-organ failure or dysfunction that would interfere with study participation
* Previous enrollment in conflicting clinical trials within the past 30 days
* Inability to comply with the medication regimen or study protocol

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Nocturia Frequency from Baseline to Week 8 | Baseline (Week 0) to Week 8
  The co-primary outcomes are: (1) Change in nocturia frequency, measured by Question 7 of the International Prostate Symptom Score (IPSS) which asks "Over the past month, how many times did you most typically get up to urinate from the time you went to bed at night until the time you got up in the morning?" (score range 0-5).

SECONDARY OUTCOMES:
Change in Sleep Quality from Baseline to Week 8 | Baseline (Week 0) to Week 8
  Change in sleep quality, measured by the Pittsburgh Sleep Quality Index (PSQI) total score (range 0-21, higher scores indicate worse sleep quality)

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital of School of Medicine, and International School of Medicine, International Institutes of Medicine，Zhejiang University, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
This is a single-center, investigator-initiated clinical trial with no external funding agreements or institutional policies requiring individual participant data sharing. The study involves a relatively modest sample size (n=136) from a specific patient population (post-prostate enucleation). As this is an early-phase evaluation of a traditional Chinese medicine combination therapy, we will focus on disseminating aggregated results through peer-reviewed publications and conference presentations. No formal data-sharing infrastructure or agreements are currently in place with external repositories. Patient privacy protection and compliance with local data governance regulations are prioritized for this initial study.